CLINICAL TRIAL: NCT03374423
Title: Radiofrequency for Chronic Post-mastectomy Pain: is it Better to Target Intercostal Nerves (T2-T5) or Their Corresponding Dorsal Root Ganglia?
Brief Title: Radiofrequency for Chronic Post-mastectomy Pain: is it Better to Target Intercostal Nerves or Corresponding Dorsal Root Ganglia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diab Fuad Hetta, clinical professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENPH
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Post-Mastectomy Chronic Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intercostal nerve group (Active Comparator): pulsed radiofrequency on intercostal nerves (2-5)
  Interventions: Procedure: radiofrequency
- dorsal root ganglion group (Active Comparator): pulsed radiofrequency on dorsal root ganglion (2-5)
  Interventions: Procedure: radiofrequency

INTERVENTIONS:
Procedure: radiofrequency — The procedure will be done under propofol sedation, under fluoroscopic guidance. The image intensifier will be rotated in a cephalo-caudal direction until the endplates of the thoracic vertebrae are aligned and the transverse processes became discernable from the ribs.
  For the intercostal nerve group, the radiofrequency needle 10 cm with 10 ml active tip will then inserted to contact the lower edge of the transverse process of (T2-T5), the needle is walked off to obtain sensory stimulation between 0.3-0.6 mv and motor stimulation less than 1.2 mv .five cycle of pulsed radiofrequency will be delivered.
  Arms: intercostal nerve group
Procedure: radiofrequency — The procedure will be done under propofol sedation, under fluoroscopic guidance.for dorsal root ganglion group, radiofrequency needle 10 cm with 10 ml active tip will inserted in a slightly medial-cephalad direction under the transverse processes, and using lateral fluoroscopic imaging, incrementally walked into the thoracic intervertebral foramen. Once correct needle position is confirmed, test stimulation will be performed at 50 Hz, during which time the needles will slightly redirected to optimize stimulation, the point of maximum stimulation will be designated to be the location of the dorsal root ganglion. five cycle of pulsed radiofrequency will be delivered.
  Arms: dorsal root ganglion group

SUMMARY:
neuropathic pain can occur following any surgical procedure on the breast ..

DETAILED DESCRIPTION:
chronic pain affects the daily lives of post-surgical breast cancer patients. many of these patients were undertreated for pain and generally obtained poor pain relief.treated patients with chronic thoracic segmental pain including patients with post-mastectomy pain syndrome by radiofrequency for dorsal root ganglion reported longterm pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic post-mastectomy pain for at least 3 months post operatively.
* patients with visual analogue scale for pain score > 4
* patients treated with more than one line of anti-neuropathic drugs.

Exclusion Criteria:

* patient refusal.
* coagulopathy.
* chest and back deformity.
* infection at the introduction site of the needle .

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
The intensity of pain | 1 month , 2 month and 3 month post-procedure
  A Visual Analogue Scale is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. For example, the intensity of pain. Operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end. The patient marks on the line the point that they feel represents their perception of their current state.The VAS score is determined by measuring in millimetres from the left handend of the line to the point that the patient marks.
  Scoring and interpretation : using a ruler, score is determined by measuring the distance(mm) on the10 cm line between the "no pain" anchor and the patient's mark ,providing a range of scores from (0_100).
  A higher score indicates greater pain intensity. the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm) .

SECONDARY OUTCOMES:
The analgesics consumption | 1 month , 2 month and 3 month post-procedure
  The change in analgesics consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Diab, Asyut, Assuit, Egypt

REFERENCES:
- [Background] Stevens PE, Dibble SL, Miaskowski C. Prevalence, characteristics, and impact of postmastectomy pain syndrome: an investigation of women's experiences. Pain. 1995 Apr;61(1):61-68. doi: 10.1016/0304-3959(94)00162-8. PMID 7644250
- [Background] Tasmuth T, von Smitten K, Hietanen P, Kataja M, Kalso E. Pain and other symptoms after different treatment modalities of breast cancer. Ann Oncol. 1995 May;6(5):453-9. doi: 10.1093/oxfordjournals.annonc.a059215. PMID 7669710
- [Background] Stolker RJ, Vervest AC, Groen GJ. The treatment of chronic thoracic segmental pain by radiofrequency percutaneous partial rhizotomy. J Neurosurg. 1994 Jun;80(6):986-92. doi: 10.3171/jns.1994.80.6.0986. PMID 8189279